CLINICAL TRIAL: NCT04171479
Title: A Retrospective Multicenter Post-Market Clinical Follow-up Registry Comparing Safety and Effectiveness Outcomes of Epicardial Cardiac Ablation Using Remote Navigation to Manual Techniques
Brief Title: RMN Versus Manual Epicardial Retrospective PMCF
Acronym: EPINAV
Status: Completed | Type: Observational
Sponsor: Stereotaxis (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-024
Record Dates: First submitted 2019-04-30; First posted 2019-11-21 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Tachycardia; Premature Ventricular Contraction
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Manual: Subjects who underwent epicardial mapping and/or ablation using a manual technique will comprise this group.
  Interventions: Device: Epicardial mapping and/or ablation
- Remote Magnetic Navigation: Subjects who underwent epicardial mapping and/or ablation using a remote magnetic technique (using Stereotaxis Niobe system) will comprise this group.
  Interventions: Device: Epicardial mapping and/or ablation

INTERVENTIONS:
Device: Epicardial mapping and/or ablation — Either catheter mapping, ablation, or mapping and ablation will be performed using an epicardial catheter approach.

SUMMARY:
Retrospective registry will compare subjects who've undergone a mapping and/or ablation procedure for either ischemic ventricular tachycardia or premature ventricular contraction using an epicardial approach with either manual or remote magnetic navigation. Subjects will be compared with regards to safety, efficacy and mortality.

DETAILED DESCRIPTION:
Up to 10 centers in the European Union will be selected to conduct the trial. Once a site is a selected, receives local Ethics Committee approval, and receives Sponsor approval to enroll, the site will begin enrollment. All subjects must meet eligibility criteria and follow protocol and ethics committee requirements regarding informed consent prior to enrollment. Once a subject is enrolled, the site may begin reviewing the subject's medical records and entering data into the electronic data capture system. Once enrollment and retrospective data entry is complete at a site, a monitoring visit will occur where source data verification will occur.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Have undergone an epicardial RF mapping and/or ablation for a ventricular tachycardia (VT) as standard of care treatment using either the Niobe MNS or a manual approach
* Index procedure was conducted between July 1, 2013-present date.

Exclusion Criteria:

* NA, all subjects who meet inclusion criteria may be enrolled.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone an epicardial cardiac mapping and ablation procedure using either manual or remote magnetic (using Stereotaxis Niobe system) guidance.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-02 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Acute Success | intra-operative
  Characterize acute success rates for both groups. Acute success for VT procedures is defined as non-inducibility of clinical VT and/or other monomorphic VT at the end of the index-procedure. Acute success for PVC procedures is defined as no recurrence and non-inducibility of culprit PVC at the end of the index-procedure.
Procedural Safety: rates of device-and procedure-related serious adverse events | 48 hours post index procedure
  Assess rates of device-and procedure-related serious adverse events in both groups.

SECONDARY OUTCOMES:
Chronic Success | 1 year post index procedure
  Characterize recurrence rates for both groups at 1 year post index procedure.
Chronic Safety: rates of device-or procedure-related serious adverse events | 1 year post index procedure
  Characterize rates of device-or procedure-related serious adverse events for both groups at 1 year post index procedure.
Mortality | 1 year post index procedure
  Assess mortality rate for both groups
Chronic Success | At last follow up visit, estimated up to 6 years post-procedure for some patients
  Characterize recurrence rates for both groups at last follow up.
Chronic Safety: rates of device-or procedure-related serious adverse events | At last follow up visit, estimated up to 6 years post-procedure for some patients
  Characterize rates of device-or procedure-related serious adverse events for both groups at last follow up.

CONTACTS AND LOCATIONS:
Locations (3):
- Na Homolce Hospital, Prague, Czechia
- Netherlands (2):
  - OLVG Hospital, Amsterdam
  - Erasmus Medical Center, Rotterdam